CLINICAL TRIAL: NCT06269692
Title: Multicenter randomiSed Trial on MAgnetic Resonance Imaging-guided implanTation of Cardioverter DEFibrillators
Brief Title: MAgnetic Resonance Imaging-guided implanTation of Cardioverter DEFibrillators
Acronym: SMART-DEF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Christian DE CHILLOU, Coordinating Investigator, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023-A01353-42
Record Dates: First submitted 2024-01-16; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Myocardial Infarction; Ventricular Tachycardia; Ventricular Fibrillation; Sudden Cardiac Death
Keywords: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction; Tachycardia, Ventricular; Ventricular Fibrillation; Death, Sudden, Cardiac | interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implantable Loop Recorder (Experimental): Patients identified at very low-risk of VT/VF randomized to be implanted with an ILR (experimental strategy). Following randomization, these patients will be followed using remote ILR monitoring.
  Interventions: Device: MRI screening; Device: Implantable Loop Recorder
- Implantable Cardioverter Defibrillator (Other): Patients identified at very low-risk of VT/VF randomized to be implanted with an ICD (reference strategy), which corresponds to the currently recommended treatment in post-MI patients with a LVEF ≤35% (European Society of Cardiology guidelines 2015) (Zeppenfeld et al., 2022).
  Interventions: Device: MRI screening; Device: Implantable Cardioverter Defibrillator

INTERVENTIONS:
Device: MRI screening — Cardiac Magnetic Resonance imaging for the quantification of the infarct intramural scar
Device: Implantable Loop Recorder — Inplantation of the Implantable Loop Recorder (ILR) for the patients assigned to the experimental group
  Arms: Implantable Loop Recorder
Device: Implantable Cardioverter Defibrillator — Inplantation of the Implantable Cardioverter Defibrillator (ICD) for the patients assigned to the control group, according to the current guidelines
  Arms: Implantable Cardioverter Defibrillator

SUMMARY:
Implantable cardioverter-defibrillators (ICD) are currently recommended for the primary prevention of sudden cardiac death (SCD) in patients with a remote (>6 weeks) myocardial infarction (MI) and a low (≤35%) left ventricular ejection fraction (LVEF).

Ventricular tachycardia (VT) and/or ventricular fibrillation (VF), which are responsible for most SCDs, result from the presence of surviving myocytes embedded within fibrotic MI-scar. The presence of these surviving myocytes, as well as their specific arrhythmic characteristics, is not captured by LVEF. Hence, the use of LVEF as a unique risk-stratifier of SCD results in a low proportion (17 to 31%) of appropriate ICD device therapy at 2 years. Consequently, most patients with a prophylactic ICD do not present VT/VF requiring ICD therapy prior to their first-ICD battery depletion. Thus, many patients are exposed to ICD complications, such as inappropriate shocks, without deriving any health benefit. Therefore, the current implantation strategy of prophylactic ICDs, based on LVEF only, needs to be improved in post-MI patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Patients with a LVEF≤35% assessed at least after a 40 to 90 days period (depending on the presence of coronary revascularization) following an index myocardial infarction;
* Left ventricular systolic impairment as defined by LVEF≤35% by any current standard technique (echocardiogram, multiple gated acquisition scan, or MRI) within 2 months;
* Able and willing to comply with all pre-, post- and follow-up testing, and requirements;
* Use of maximum tolerated doses of ACE inhibitors (or Angiotensin II Receptor Blockers if intolerant of ACE) and Beta Blockers and MRA as per ESC guidelines;
* Person affiliated to or beneficiary of a social security plan
* Person informed about study organization and having signed the informed consent

Exclusion Criteria:

* History of cardiac arrest or sustained VT or VF unless within 48 hours of an acute myocardial infarction;
* Standard contraindications for cardiac LGE-MRI;
* Hypersensitivity to gadolinium-based contrast agent;
* Currently implanted permanent pacemaker and/or ICD;
* Patient refusal of ICD/ILR implantation;
* Currently implanted permanent pacemaker and/or ICD;
* Clinical indication for or Cardiac Resynchronization Therapy (CRT);
* Severe renal insufficiency defined by a glomerular filtration rate (GFR) < 30 mL/min/1.73m²;
* Recent PTCA (within 30 days) or CABG (within 90 days);
* Baseline NYHA functional class IV;
* Contraindication for ICD implantation according to current guidelines;
* Woman of childbearing age without effective contraception;
* Person referred in articles L.1121-5, L. 1121-7 and L.1121-8 of the French Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1812 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2030-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Sudden Cardiac Death (SCD) during the follow-up period | 72 months
  Occurrence of SCD during the follow-up period, as defined by the World Health Organization in 10-ICD: death occurring within 24 hours from onset of symptoms.

SECONDARY OUTCOMES:
Total number of deaths during the follow-up period | 72 months
Total number of deaths from cardiovascular cause during the follow-up period | 72 months
Total number of SCD due to ventricular arrhythmia during the follow-up period | 72 months
Total number (per patient) of sustained VT episodes treated by the ICD or recorded by the ILR during the follow-up period | 72 months
Total number (per patient) of VF episodes treated by the ICD or recorded by the ILR during the follow-up period | 72 months
Total number of hospitalizations due to cardiovascular causes during the follow-up period | 72 months
Duration of hospitalizations due to cardiovascular causes during the follow-up period | 72 months
Total number of hospitalizations from any cause during the follow-up period | 72 months
Duration of hospitalizations from any cause during the follow-up period | 72 months
Quality of life assessed by the scoring obtained from EuroQol questionnaires (EQ-5D-5L) during the follow-up period | 72 months
Measurements of the estimated costs | 72 months
  Measurements of the estimated costs for the National Health Insurance System (NHIS) in the different arms of the trial
Dice scores of the segmentation of the left ventricle and scar obtained from new MR sequences | 36 months
  Dice scores of the segmentation of the left ventricle and scar obtained from new MR sequences, LGE segmentation by cardiologists/radiologists as the ground truth
Contour distance metrics of the segmentation of the left ventricle and scar obtained from new MR sequences | 36 months
  Contour distance metrics of the segmentation of the left ventricle and scar obtained from new MR sequences, LGE segmentation by cardiologists/radiologists as the ground truth
Dice scores of the accuracy of fully automated segmentation of the left ventricle and scar | 36 months
  Dice scores of the accuracy of fully automated segmentation of the left ventricle and scar, using manually corrected segmentation by cardiologists/radiologists as the ground truth
Contour distance metrics of the accuracy of fully automated segmentation of the left ventricle and scar | 36 months
  Contour distance metrics of the accuracy of fully automated segmentation of the left ventricle and scar, using manually corrected segmentation by cardiologists/radiologists as the ground truth

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No